CLINICAL TRIAL: NCT01994772
Title: Therapeutic Hypothermia After Cardiac Arrest in Non Shockable Rhythm at Rescue Arrival: The HYPERION Study
Brief Title: Therapeutic Hypothermia After Cardiac Arrest in Non Shockable Rhythm
Acronym: HYPERION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RCB 2012-A00405-38
Record Dates: First submitted 2013-11-07; First posted 2013-11-26 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Arrest
Keywords: Therapeutic hypothermia; Targeted controlled temperature; Cardiac arrest; Non shockable rhythm; successful resuscitation
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted controlled temperature between 32.5 and 33.5°C (Active Comparator): Patients will be placed in targeted temperature control between 32.5 and 33.5 ° C for 24 hours and then slowly rewarmed for targeted temperature control between 36.5 and 37.5 ° C for 24 hours.
  Interventions: Procedure: Targeted controlled temperature between 32.5 and 33.5°C; Procedure: Targeted controlled temperature between 36.5 and 37.5°C
- Targeted controlled temperature between 36.5 and 37.5°C (Placebo Comparator): Patients will be placed in targeted temperature control between 36.5 and 37.5 ° C for 48 hours.
  Interventions: Procedure: Targeted controlled temperature between 36.5 and 37.5°C

INTERVENTIONS:
Procedure: Targeted controlled temperature between 32.5 and 33.5°C — Therapeutic hypothermia ie targeted controlled temperature between 32.5° and 33.5°C will be induced in the active group. Usual method of controlled temperature will be use in ICU: internal active method or external active method.
  Other Names: Therapeutic hypothermia; Induce hypothermia
  Arms: Targeted controlled temperature between 32.5 and 33.5°C
Procedure: Targeted controlled temperature between 36.5 and 37.5°C — Temperature was maintain between 36.5° and 37.5°C in the control group. In case of temperature superior to 37.5°C or inferior to 36.5°C, a pharmaceutical treatment and/or active cooling or warming was introduce to maintain temperature between the range of 36.5 - 37.5°C.
  Other Names: Normothermia

SUMMARY:
Cardiac arrest is at present a major cause of mortality as well as a cause of disability for the surviving victims.In Europe, every year counts as 300,000 cardiac arrests responsible for 250,000 deaths. Thus, less than 20 % of patients discharged home with impaired quality of life associated with symptoms of tiredness, stress, anxiety. The prognosis is related to the initial cardiac rhythm present during the initiation of resuscitation. Recent progress in the improvement of mortality and neurological outcome has been achieved over the last decade thanks to the systematic implementation of a period of targeted temperature control between 32 and 34 ° C in patients who benefited from the realization of at least one electrical external shock.

There are theoretical and clinical arguments to think that achieving the same way a period of targeted temperature control between 32 and 34 ° C in patients treated for cardiac arrest with a non- shockable rhythm on arrival can also benefit from this procedure. However other arguments are against this hypothesis including an increase in the risk of infection , worsening of the patient's hemodynamic status with no benefit to him. To answer this question, we conduce a randomized multicenter study testing the potential improvement of neurological outcome through this procedure targeted temperature control between 32.5 and 33.5 ° C in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest in non shockable rhythm
* Glasgow score ≤ 8

Exclusion Criteria:

* No flow > 10 min
* Low flow > 60 min
* Major hemodynamic instability
* Delay between cardiac arrest and inclusion > 300 min
* Cirrhosis Child C
* Age < 18 years
* Pregnant women
* Patient with no liberty
* Lack of informed consent
* Prior inclusion in a research protocol involving cardiac arrest with draw, and whose primary endpoint focuses on the evaluation of a neurological score Day 90

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2014-01-26 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Neurological outcome assessed with Cerebral Performance Category scale | Day 90

SECONDARY OUTCOMES:
Intensive Care Unit Mortality | Discharge from Intensive Care Unit, an expected average of 7 days
  Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 7 days.
Hospital Mortality | Discharge from hospital, an expected average of 2 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Mortality at day 90 | Day 90
Quality of life Score | Day 90
  Quality of life at day 90 will be assessed by 36-Items Short Form for Health Survey telephonic interview
Life autonomy | Day 90
  Life autonomy will be assessed by Index Activity of Daily Living, modified Barthel index, and by two normative question about life autonomy
Neurocognitive evaluation | Day 90
  Neurocognitive status will be assessed by telephonic validated version of Mini Mental State Examination
Post traumatic stress disorders symptoms | Day 90
  Post traumatic stress disorders symptoms will be assessed by Impact Event Scale Revised
Intensive Care Unit length of stay | Discharge from Intensive Care Unit, an expected average of 7 days
  Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 7 days
Hospital length of stay | Discharge from hospital, an expected average of 2 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Mechanical ventilation duration | Time from extubation, an expected average of 4 days
  Participants will be followed for the duration of mechanical ventilation, an expected average of 4 days
Severe hemorrhage | Intensive care unit length of stay, an expected average of 7 days
  Severe hemorrhage is define by transfusion of 1 or more blood product requirement and/or intracranial hemorrhage. Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days.
Nosocomial Bloodstream infection | Intensive care unit length of stay, an expected average of 7 days
  Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days.
Early onset pneumonia | 2 days
Ventilated Associated Pneumonia | Duration of mechanical ventilation, an expected average of 4 days
  Participants will be followed for the duration of mechanical ventilation, an expected average of 4 days
Central Veinous Catheter infection | Intensive care unit length of stay, an expected average of 7 days
  Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days.
Total dose of inotropic drugs | 48 hours
  Total dose of different inotropic drugs (Epinephrine, Norepinephrine, Dobutamine) will be compare between 2 groups during targetted controlled temperature management period.
Extra renal support requirement | Intensive care unit length of stay, an expected 7 days
  Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days
Acute pulmonary oedema by left ventricular failure | Intensive care length of stay, an expected 7 days
  Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days.
Seizure | Intensive care length of stay, an expected 7 days
  Participants will be followed for the duration of Intensive care unit stay, an expected average of 7 days
Severe arrythmia | Intensive care unit length of stay, an expected 7 days
  Severe arrythmia will be define by salvo of ventricular extrasystole, ventricular fibrillation, ventricular tachycardia, need an external shock, need anti-arrhythmic treatment. Participants will be followed for the duration of Intensive Care Unit stay, an expected average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste Lascarrou, MD, Study Chair — Nantes University Hospital
Locations (26):
- France (25):
  - Medical Intensive Care Unit, Angers
  - Medical Surgical Intensive Care Unit, Angoulême
  - Medical Intensive Care Unit, Annecy
  - Medical Surgical Intensive Care Unit, Argenteuil
  - Medical Intensive Care Unit, Clermont-Ferrand
  - Medical Intensive Care Unit, Dijon
  - Medical Surgical Intensive Care Unit, La Roche-sur-Yon
  - Medical Surgical Intensive Care Unit, Le Mans
  - Medical Surgical Intensive Care Unit, Lens
  - Medical Intensive Care Unit, Lille
  - Medical Surgical Intensive Care Unit, Limoges
  - Medical Surgical Intensive Care Unit, Lorient
  - Medical Surgical Intensive Care Unit, Montauban
  - Medical Intensive Care Unit, Nantes
  - Medical Intensive Care Unit, Orléans
  - Cochin University Hospital Center, Paris
  - Medical Intensive Care Unit, Poitiers
  - Medical Surgical Intensive Care Unit, Roanne
  - Medical Surgical Intensive Care Unit, Rodez
  - Medical Surgical Intensive Care Unit, Saint-Brieuc
  - Medical Surgical Intensive Care Unit, Saint-Nazaire
  - Medical Surgical Intensive Care Unit, St-Malo
  - Medical Intensive Care Unit, Strasbourg
  - Medical Intensive Care Unit, Tours
  - Medical Surgical Intensive Care Unit, Versailles
- CHU Pointe à Pitre, Pointe-à-Pitre, Guadeloupe

REFERENCES:
- [Derived] Lascarrou JB, Ermel C, Cariou A, Laitio T, Kirkegaard H, Soreide E, Grejs AM, Reinikainen M, Colin G, Taccone FS, Le Gouge A, Skrifvars MB. Dysnatremia at ICU admission and functional outcome of cardiac arrest: insights from four randomised controlled trials. Crit Care. 2023 Dec 1;27(1):472. doi: 10.1186/s13054-023-04715-z. PMID 38041177
- [Derived] Ziriat I, Le Thuaut A, Colin G, Merdji H, Grillet G, Girardie P, Souweine B, Dequin PF, Boulain T, Frat JP, Asfar P, Francois B, Landais M, Plantefeve G, Quenot JP, Chakarian JC, Sirodot M, Legriel S, Massart N, Thevenin D, Desachy A, Delahaye A, Botoc V, Vimeux S, Martino F, Reignier J, Cariou A, Lascarrou JB. Outcomes of mild-to-moderate postresuscitation shock after non-shockable cardiac arrest and association with temperature management: a post hoc analysis of HYPERION trial data. Ann Intensive Care. 2022 Oct 17;12(1):96. doi: 10.1186/s13613-022-01071-z. PMID 36251223
- [Derived] Lascarrou JB, Merdji H, Le Gouge A, Colin G, Grillet G, Girardie P, Coupez E, Dequin PF, Cariou A, Boulain T, Brule N, Frat JP, Asfar P, Pichon N, Landais M, Plantefeve G, Quenot JP, Chakarian JC, Sirodot M, Legriel S, Letheulle J, Thevenin D, Desachy A, Delahaye A, Botoc V, Vimeux S, Martino F, Giraudeau B, Reignier J; CRICS-TRIGGERSEP Group. Targeted Temperature Management for Cardiac Arrest with Nonshockable Rhythm. N Engl J Med. 2019 Dec 12;381(24):2327-2337. doi: 10.1056/NEJMoa1906661. Epub 2019 Oct 2. PMID 31577396
- [Derived] Lascarrou JB, Meziani F, Le Gouge A, Boulain T, Bousser J, Belliard G, Asfar P, Frat JP, Dequin PF, Gouello JP, Delahaye A, Hssain AA, Chakarian JC, Pichon N, Desachy A, Bellec F, Thevenin D, Quenot JP, Sirodot M, Labadie F, Plantefeve G, Vivier D, Girardie P, Giraudeau B, Reignier J; Clinical Research in Intensive Care and Sepsis (CRICS) Group and HYPERION Study Group. Therapeutic hypothermia after nonshockable cardiac arrest: the HYPERION multicenter, randomized, controlled, assessor-blinded, superiority trial. Scand J Trauma Resusc Emerg Med. 2015 Mar 7;23:26. doi: 10.1186/s13049-015-0103-5. PMID 25882712
- See also: Related Info — http://www.sjtrem.com/content/23/1/26